CLINICAL TRIAL: NCT03905083
Title: miRNA and Myokines Acutely-expressed During Exercise in Patients With Pulmonary Arterial Hypertension
Brief Title: miRNA and Myokines in Patients With PAH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics related to research activity
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Michael Risbano, Head, Clinical Operations for Pulmonary Hypertension, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY19120032
Record Dates: First submitted 2019-02-25; First posted 2019-04-05 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2021-02

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise rehab (Experimental): Investigators aim to evaluate how exercise training may provide beneficial effects on the skeletal muscle and/or pulmonary vasculature in select subjects with pulmonary arterial hypertension, scleroderma or mixed connective tissue disease or patients with exercise pulmonary arterial hypertension
  Interventions: Other: Exercise Rehab
- No exercsie rehab (No Intervention): Some participants will not be assigned to do exercise rehab so we would be using them as a control arm to intervention group

INTERVENTIONS:
Other: Exercise Rehab — Participants who do the Exercise Rehab will engage in up to four center-based exercise rehab sessions each week for approximately 12 weeks; each session lasting roughly 1-hour with a stimulus (exercise) phase and a mix of warm up and cool down. Cycle ergometer and treadmill exercise may be used.
  Arms: Exercise rehab

SUMMARY:
The overall objective of this study is to fulfill the Pilot study (miRNA and Myokines Acutely-expressed During Exercise) goal to Investigate the excretion of skeletal muscle-derived miRNA and myokines in patients with pulmonary arterial hypertension during acute exercise that are biologically active and modulate skeletal muscle function during exercise.

Pulmonary arterial hypertension (PAH), is characterized by the proliferation of endothelial and smooth muscle cells within the precapillary pulmonary vasculature, if untreated results in increased pulmonary vascular resistance and death. The hallmark perivascular infiltrates in PAH contain inflammatory macrophages and lymphocytes resulting in endothelial dysfunction and involves the dysregulation of distinct inflammatory mechanisms. Idiopathic PAH (iPAH) and scleroderma-associated PAH (SSc-PAH), are related by similar clinical and pathophysiologic features. Patients with PAH experience a central cardiovascular limitation to exercise. Despite effective treatment with pulmonary vasodilators, many resting PAH (rPAH) patients continue to experience exercise intolerance. PAH is increasingly acknowledged as a systemic disease, beyond abnormalities of the pulmonary vasculature. Although other contributions to exercise intolerance in PAH exist, skeletal muscle dysfunction significantly impacts exercise tolerance. The molecular mechanisms behind skeletal muscle dysfunction in PAH remain unclear. Provocative testing with invasive cardiopulmonary exercise testing challenges the cardio-pulmonary-vascular and skeletal muscle systems and elicits a cascade of physiologic events not measurable at rest. Myokines are circulating mediators released from skeletal muscle in an endocrine-like fashion in disease and health influencing many factors but not limited to systemic inflammation, immunity and endothelial function. Myokines have not been well described in PAH. Preliminary data indicate that myokines play important, yet still undescribed, roles in this disease. MicroRNAs (miRNAs) are small non-coding RNA molecules, which negatively regulate gene expression via repressing translation and degrading messenger RNAs through sequence-specific binding. There is a growing literature regarding the biological activity of extracellular miRNAs in PAH and in aerobic exercise. miR-126 has been implicated in skeletal muscle dysfunction in PAH, while miR-133 is skeletal muscle-specific but unlike miR-126 it is not yet implicated in skeletal muscle dysfunction in PAH.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a RHC/iCPET procedure at the UPMC Presbyterian Hospital Catheterization Lab.
* 18 years of age or older
* Able to read and understand the informed consent.
* Subjects who have signed the iCPET registry consent.

Exclusion Criteria:

* Pregnant women
* people under 18
* Who are unable to read and understand the informed consent.
* Subjects prescribed anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of released miRNA/myokines on the skeletal muscle in PAH patients. | At the time of the procedure
  We will be able to measure the levels of miRNA by doing RNA sequencing and then To evaluate the impact of released miRNA/myokines on the skeletal muscle in PAH patients.Protein and transcript levels will be confirmed using Western blots and real-time PCR
To evaluate the impact of formal exercise training on the skeletal muscle | At the time of the procedure
  Muscle biopsy for miRNA and myokine assessment will be performed for this outcome. Total RNA and protein extracted from quadriceps muscle biopsies will be used to measure RNA and protein expression. We will perform a secretome analysis utilizing the Mass Spectrometry Lab at the University of Pittsburgh for an unbiased assessment of muscle-secreted myokines in our subjects.
  RNA sequencing and then Protein and transcript levels will be confirmed using Western blots and real-time PCR
To evaluate the impact of formal exercise training on the pulmonary vasculature system | At the time of the procedure
  This will be done by measuring hemodynamics during invasive cardiopulmonary exercise test. We will correlate miRNA and myokines released from the skeletal muscle with measures of oxygen delivery and extraction in the muscle and oxygen consumption - calculated from arterial and pulmonary artery blood gasses and invasive hemodynamics. Oxygen delivery to peripheral tissues is determined by (Q ) ̇x CaO2. Oxygen extraction is Ca-vO2. Oxygen consumption is continuously measured by iCPET as( V) ̇O2. Systemic oxygen extraction ratio is determined by (Ca-vO2)/ CaO2

CONTACTS AND LOCATIONS:
Overall Officials: Michael Risbano, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Division of Pulmonary, Allergy and Critical Care Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Our IPD plan would include:
  1. The use of a controlled access approach, using a transparent and robust system to review requests and provide secure data access through asking data requester to fill up formal application that would give details on how this data would be used.
  2. Seeking consent for sharing IPD from the clinical trial participants with adequate assurance that patient privacy and confidentiality can be maintained.
  3. Establishing an approach to resource the sharing of IPD which would include support from trial funders, sponsor organizations and users of IPD.